CLINICAL TRIAL: NCT00758459
Title: A 6 Week Double-Blind, Placebo-controlled, Randomised, Parallel Group Phase IIa Study to Assess the Tolerability/Safety and Efficacy of AZD1236as an Oral Tablet in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Safety/Tolerability Study With AZD1236 in Chronic Obstructive Pulmonary Disease (COPD) Patients
Acronym: CERA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Andrew Lockton, MD, Medical Science Director, Emerging Products, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D4260C00003
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2011-08-19 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — 4-((5-chloro-2-pyridinyl)oxy)-1-((((4S)-4-methyl-2,5-dioxo-4-imidazolidinyl)methyl)sulfonyl)-piperidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD1236
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1236 — oral tablet, 75 mg, twice daily during 6 weeks
  Arms: 1
Drug: Placebo — Dosing to match AZD1236
  Arms: 2

SUMMARY:
The primary aim of this study is to investigate the tolerability and safety of AZD 1236 compared with placebo ("inactive substance") in COPD patients by assessment of Adverse Events, vital signs and laboratory safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD for 1 month
* Men or postmenopausal women
* Spirometry values indicating reduced lung function
* Smoking history equivalent to using 20 cigarettes a day for 10 years

Exclusion Criteria:

* Any current respiratory tract disorders other than COPD
* Requirement for regular oxygen therapy
* Use of oral or parenteral glucocorticosteroids within 30 days prior to the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-09; Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helgo Magnussen, MD, Professor, Principal Investigator — Pulmonary research institute at Hospital Grosshansdorf, Wöhrendamm, Grosshansdorf Germany; Andrew Lockton, MD, Study Director — AstraZeneca R&D Charnwood
Locations (14):
- Bulgaria (2):
  - Research Site, Rousse
  - Research Site, Sofia
- Finland (3):
  - Research Site, Helsinki
  - Research Site, Oulu
  - Research Site, Preitilä
- Germany (2):
  - Research Site, Berlin
  - Research Site, Grobhansdorf
- Hungary (4):
  - Research Site, Győr
  - Research Site, Komló
  - Research Site, Pécs
  - Research Site, Vásárosnamény
- Slovakia (3):
  - Research Site, Bojnice
  - Research Site, Liptovský Hrádok
  - Research Site, Žilina

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD1236: AZD1236
- Placebo: Placebo
Period: Overall Study
Arm/Group | AZD1236 | Placebo
Started | 35 | 39
Completed | 32 | 35
Not Completed | 3 | 4
Not completed — Adverse Event | 3 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1236 | Placebo | Total
Number analyzed (Participants) | 35 | 39 | 74
Age Continuous [Mean (Full Range); unit: Year] | 61.7 [48 to 76] | 61.7 [46 to 77] | 61.7 [46 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 24 | 27 | 51

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: Number of patients who had an Adverse Event
Time Frame: all study visits
Measure: Number; unit: Participants
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 35 | 39
Participants | 13 | 17

2. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Change in FEV1 from baseline to end of treatment
Time Frame: Before treatment and after 1, 2, 4 and 6 weeks of treatment
Measure: Mean (Full Range); unit: L
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 35 | 39
L | -0.006 (-0.410) [-0.410 to 0.450] | 0.003 (-0.450) [-0.450 to 0.990]

3. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Change in FVC from baseline to end of treatment
Time Frame: Before treatment and after 1, 2, 4 and 6 weeks of treatment
Measure: Mean (Full Range); unit: L
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 35 | 39
L | -0.048 (-0.760) [-0.760 to 0.660] | -0.028 (-0.730) [-0.730 to 0.940]

4. Secondary Outcome: Vital Capacity (VC)
Description: Change in VC from baseline to end of treatment
Time Frame: Before treatment and after 1, 2, 4 and 6 weeks of treatment
Measure: Mean (Full Range); unit: L
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 35 | 39
L | -0.025 (-0.840) [-0.840 to 0.660] | -0.043 (-1.03) [-1.03 to 1.09]

5. Secondary Outcome: Inspiratory Capacity (IC)
Description: Change in IC from baseline to end of treatment
Time Frame: Before treatment and after 1, 2, 4 and 6 weeks of treatment
Measure: Mean (Full Range); unit: L
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 35 | 39
L | -0.083 (-0.730) [-0.730 to 0.720] | 0.053 (-0.620) [-0.620 to 1.55]

6. Secondary Outcome: Forced Expiratory Flow (FEF)25-75%
Description: Change in FEF from baseline to end of treatment
Time Frame: Before treatment and after 1, 2, 4 and 6 weeks of treatment
Measure: Mean (Full Range); unit: L/s
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 35 | 39
L/s | -0.073 (-1.45) [-1.45 to 0.250] | 0.010 (-0.280) [-0.280 to 1.06]

7. Secondary Outcome: Peak Expiratory Flow (PEF) Morning
Description: Change in PEF from average during run-in to average during the last 4 w of treatment
Time Frame: Daily during run-in and treatment
Measure: Mean (Full Range); unit: L/min
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 35 | 39
L/min | 1.45 (-78.4) [-78.4 to 71.5] | 7.47 (-57.0) [-57.0 to 138]

8. Secondary Outcome: Peak Expiratory Flow (PEF) Evening
Description: Change in PEF from average during run-in to average during the last 4 w of treatment
Time Frame: Daily during run-in and treatment
Measure: Mean (Full Range); unit: L/min
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 35 | 39
L/min | 7.48 (-70.4) [-70.4 to 79.6] | 6.69 (-48.1) [-48.1 to 139]

9. Secondary Outcome: Clinical Chronic Obstructive Pulmonary Disease (COPD) Questionnaire(CCQ) Total
Description: Change from baseline to end of treatment in score , The total scores vary between 0 (never/not limited at all) to 6 (almost all the time/totally limited)
Time Frame: Before treatment and after 1, 2, 4 and 6 weeks of treatment
Measure: Mean (Full Range); unit: Score on scale
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 35 | 39
Score on scale | 0.373 (0.270) [0.270 to 0.900] | -0.374 (-4.80) [-4.80 to 1.30]

10. Secondary Outcome: Clinical Chronic Obstructive Pulmonary Disease (COPD) Symptoms, Breathlessness
Description: Change in COPD symptom, Breathlessness from average during run-in to average during the last 4 w of treatment. 5-point Likert-type scale, ranging from 0 (none) to 4 (severe)
Time Frame: Daily during run-in and treatment
Measure: Mean (Full Range); unit: Score on scale
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 35 | 39
Score on scale | -0.173 (-1.22) [-1.22 to 0.885] | -0.390 (-2.15) [-2.15 to 0.567]

11. Secondary Outcome: Clinical Chronic Obstructive Pulmonary Disease (COPD) Symptoms, Chest Tightness
Description: Change in COPD symptom, chest tightness from average during run-in to average during the last 4 w of treatment, 5-point Likert-type scale, ranging from 0 (none) to 4 (severe)
Time Frame: Daily during run-in and treatment
Measure: Mean (Full Range); unit: Scores on a Scale
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 35 | 39
Scores on a Scale | -0.073 (-1.10) [-1.10 to 1.28] | -0.212 (-1.89) [-1.89 to 1.41]

12. Secondary Outcome: Clinical Chronic Obstructive Pulmonary Disease (COPD) Symptoms, Cough Score
Description: Change in COPD symptoms, cough score from average during run-in to average during the last 4 w of treatment, 5-point Likert-type scale, ranging from 0 (none) to 4 (severe)
Time Frame: Daily during run-in and treatment
Measure: Mean (Full Range); unit: Scores on a Scale
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 35 | 39
Scores on a Scale | -0.200 (-1.36) [-1.36 to 1.53] | -0.470 (-1.73) [-1.73 to 0.752]

13. Secondary Outcome: Clinical Chronic Obstructive Pulmonary Disease (COPD) Symptoms, Night Time Awakenings
Description: Change in night time awakenings from average during run-in to average during the last 4 w of treatment, 5-point Likert-type scale, ranging from 0 (none) to 4 (severe)
Time Frame: Daily during run-in and treatment
Measure: Mean (Full Range); unit: Score on scale
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 35 | 39
Score on scale | -0.128 (-1.11) [-1.11 to 1.03] | -0.262 (-2.00) [-2.00 to 0.852]

14. Secondary Outcome: 6-minute Walk Test
Description: Change from baseline to end of treatment
Time Frame: Before treatment and after 6 weeks of treatment
Measure: Mean (Full Range); unit: m
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 35 | 39
m | 14.4 (-117) [-117 to 200] | 9.68 (-111) [-111 to 150]

ADVERSE EVENTS:
Arm/Group | AZD1236 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/39
Other Adverse Events (participants affected / at risk) | 8/35 | 8/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1236 (N=35) | Placebo (N=39)
Pharyngeal Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1236 (N=35) | Placebo (N=39)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 3 | 4
HEADACHE (Nervous system disorders) | 4 | 1
VIRAL INFECTION (Infections and infestations) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less